CLINICAL TRIAL: NCT07350395
Title: Assessing the Impact of Glucocorticoids in Children and Young People With Rheumatic Conditions, to Develop a Patient Reported Outcome Measure (PROM).
Brief Title: Exploring and Measuring the Impact of Steroids in Children and Young People
Status: Recruiting | Type: Observational
Sponsor: University of the West of England (Other)
Collaborators: Alder Hey Children's NHS Foundation Trust (Other); Bristol Royal Hospital for Children (Other); Glasgow Royal Hospital for children (Unknown)
Responsible Party: Sponsor
Other Study IDs: 352096
Record Dates: First submitted 2025-09-23; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Rheumatic Diseases; Rheumatic Disorder; Rheumatologic Conditions (JRA,Lupus)
Keywords: rheumatic diseases; children and young people; steroids; glucocorticoids; qualitative
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Focus groups for parents with children under 8 years old
- Focus groups with children 8-12 years old
- Focus groups for young people aged 13-15 years old
- Focus groups for young people aged 16-18 years old
- Cognitive interviewing for parents with children under 8 years old
- Cognitive interviewing for children 8-12 years old
- Cognitive interviewing for young people aged 16-18 years old
- Cognitive interviewing for young people aged 13-15 years old

SUMMARY:
Assessing the impact of glucocorticoids in children and young people with rheumatic conditions, to develop a patient reported outcome measure (PROM).

Glucocorticoids, also known as steroids, are a very effective medication for the treatment of rheumatological conditions. They are used to reduce inflammation, pain and damage to organs. However, steroids can have some unwanted side effects, such as, increased weight, skin changes, feeling anxious, delayed puberty, diabetes and loss of bone mass. These side effects can therefore impact children and young people's health related quality of life (HRQoL).

The investigators would like to create a new questionnaire for children and young people (CYP) who take steroids due to their rheumatological condition. The questionnaire, called a Patient Reported Outcome Measure, (PROM), will measure how steroids are affecting CYP. The first step in creating the questionnaire is to talk to children, young people and their parents/guardians about their experiences of taking steroids. The investigators plan to do this in focus groups, with people around the same age. The second step will then be to take everything people said in the focus group to create the questions in the questionnaire. Cognitive interviewing will then be used in a structured one on one interview to test for relevance, clarity and understanding of the questions.

Children, young people and their parents/guardians will be involved throughout the research. Children and young people will give their thoughts and feedback on resources created for participants (consent forms/assent forms/participation information sheet/interview schedule), as well as how the focus groups and cognitive interviews should be structured.

With consent, participants will be provided with a lay summary of the results. Results will also be published within peer-reviewed journals, special interest groups, trial meetings, patient charity meetings and presented at conferences.

ELIGIBILITY:
Inclusion Criteria:

* 1. Rheumatology patients aged 0 to18 years old. 2. Patients should have capacity to assent or consent immediately prior to the interview.

  3. The patient should have a good understanding of spoken and written English be able to understand the participant information sheets, assent/consent forms.

  4. Treatment with glucocorticoids with intravenous or oral glucocorticoids for an autoimmune or inflammatory condition within the previous two years (or longer duration).

Parents/guardians:

1. Parents (mother/ father) or legal guardians of rheumatological patients fulfilling criteria 1-4 above.
2. Parents or legal guardians should have capacity to consent for themselves (+/- their child) immediately prior to the interview.
3. The parents or legal guardians should have a good understanding of spoken and written English be able to understand the participant information sheets, assent/consent forms.

Exclusion Criteria:

* 1. Rheumatology patients who are more than 18 years of age. 2. Patients who do not have capacity to assent or consent immediately prior to the interview.

  3. Patient who have insufficient understanding of spoken and written English be able to understand the participant information sheets, assent/consent forms.

  4. Patients who either have never taken steroids or have not taken steroids within the last two years as part of their treatment plan for their rheumatological condition.

  5. Relative is not a parent or legal guardian. 6. Parents/guardians of rheumatology patients fulfilling any of the exclusion criteria above.

  7. Parents/guardians who do not have capacity to assent or consent immediately prior to the interview.

  8. Parents/guardians who have insufficient understanding of spoken and written English be able to understand the participant information sheets, assent/consent forms.

  9. Parents/guardians of rheumatology patients who have never taken steroids or have not taken steroids within the last two years as part of their treatment plan for their rheumatological condition.

  10. Membership of the steering committee

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Three NHS sites (paediatric rheumatology clinics) will be used for recruitment of participants:
  Bristol Royal Hospital for Children Alder Hey Children's Hospital (Liverpool) Royal Hospital for Children (Glasgow)
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To explore the impact of glucocorticoids (steroids) on health-related quality of life (HRQoL) in CYP. | Through study completion, an average of 1 year.
  To develop a long list of potential questionnaire items for one or more patient reported outcome measures (PRO) for children and young people, who are treated with glucocorticoids, which assesses its impact of this treatment on their symptoms and everyday life.

SECONDARY OUTCOMES:
Secondary analysis of specific topics of greatest importance to patients and families may be performed based on anonymised qualitative dataset from objective 1 | Through study completion, an average of 1 year.
  Secondary analyses may in future also be used to explore specific topics of importance within the qualitative data, depending on what emerges as of greatest importance (e.g. impact on appearance, sense of self).

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Bristol Royal Hospital for Children, Bristol, North Somerset
  - Royal Hospital for children Glasgow, Glasgow, North Somerset
  - Alder Hey Hospital, Liverpool, North Somerset

IPD SHARING:
Plan to Share IPD: Undecided
This is not a trial, it is an exploratory qualitative study, therefore outcome measures are not relevant.